CLINICAL TRIAL: NCT03351270
Title: Prospective, Longitudinal Study of the Natural History and Functional Status of Patients With Myotubular Myopathy and Other CentroNuclear Myopathies
Brief Title: Prospective Natural History Study of Patients With Myotubular Myopathy and Other CentroNuclear Myopathies
Acronym: NatHis-CNM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Myologie, France (Other)
Collaborators: Dynacure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NatHis-CNM
Record Dates: First submitted 2017-11-14; First posted 2017-11-22 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Centronuclear Myopathy
Keywords: CNM; XLMTM; Myotubular myopathy
MeSH Terms: conditions — Myopathies, Structural, Congenital | interventions — Respiratory Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Standardized strength, respiratory and motor function assessments — Standardized assessments will be adjusted by the age, the ambulant status and the respiratory status of the patient. The visit frequency will also be adjusted according to the age and to the time spent in the study varying between quarterly to yearly.

SUMMARY:
This is the 2 years extension of the prospective and longitudinal study of the natural history and functional status of patients with myotubular myopathy and other centronuclear (CNM) sponsored by Dynacure including ten additional pediatric patients with mutation in MTM1 or DNM2 genes). the patients are planned to be enrolled in one year leading to an expected total number of 70 patients followed at least over 1 year period. Data from the study will be used to characterize the disease course of CNM and determine which outcome measures will be the best to assess the efficacy of potential therapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age (newborns included) may participate
* Patients over 18 years of age and parent(s)/legal guardian(s) of patients < 18 years of age must be provide written informed consent prior to participating in the study and informed assent will be obtained from minors at least 7 years of age when required by regulation.
* Myotubular Centronuclear myopathy (MTMCNM) resulting from a mutation in the MTM1, DNM2 or BIN1 gene
* Male or symptomatic female. A symptomatic female will be defined by the motor function assessment by Motor Function Measure (MFM) or North Star Ambulatory Assessment (NSAA) below 80% of the total score.
* Willing and able to comply with all protocol requirements and procedures.
* In France only: Affiliated to or a beneficiary of a social security category

Exclusion Criteria:

* Other disease which may significantly interfere with the assessment of the MTM CNM and is clearly not related to the disease
* Currently enrolled in a treatment study; or treatment with an experimental therapy other than pyridostigmine
* For women: pregnancy or current breastfeeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-28 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
MFM score change from baseline | Baseline, 6 months, 12 months and every year up to 60 months
  Motor Function Measure scale. The total test score can range from 0 if the subject cannot perform any of the items to 100 if all the items are fully achieved.
CHOP-INTEND score change from baseline | Baseline, 6 months, 12 months and every year up to 60 months
  Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders
Modified Hammersmith score change from baseline | Baseline, 6 months, 12 months and every year up to 60 months
  Modified Hammersmith Functional Motor Scale. The total test score can range from 0 if the subject cannot perform any of the items to 40 if all the items are fully achieved
Moviplate score change from baseline | Baseline, 6 months, 12 months and every year up to 60 months
  Moviplate score
6MWD change from baseline | Baseline, 6 months, 12 months and every year up to 60 months
  6 Minute Walking Distance
Grip strength change from baseline | Baseline, 6 months, 12 months and every year up to 60 months
  MyoGrip
Pinch strength change from baseline | Baseline, 6 months, 12 months and every year up to 60 months
  MyoPinch
Forced Vital Capacity change from baseline | Baseline, 6 months, 12 months and every year up to 60 months
Peak Cough Flow change from baseline | Baseline, 6 months, 12 months and every year up to 60 months
Maximum Inspiratory Pressure change from baseline | Baseline, 6 months, 12 months and every year up to 60 months
Maximum Expiratory Pressure change from baseline | Baseline, 6 months, 12 months and every year up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Servais, MD, Principal Investigator — Centre de référence neuromusculaire, CHR La Citadelle; 4000 Liege Belgium
Locations (11):
- Centre de référence neuromusculaire, CHR La Citadelle, Liège, Belgium
- France (7):
  - Hôpital Femme Mère Enfant, CHU Lyon L'Escale, Bron
  - Hôpital Roger Salengro, CHU Lille, Lille
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital Armand Trousseau, Paris
  - I-Motion Institute - Trousseau Hospital, Paris
  - Institute of Myology, Paris
  - Hôpital Sainte Musse, Toulon
- Universitätsklinikum Essen (AöR), Essen, Germany
- Bambino Gesu Children's Hospital, Roma, Italy
- Hospital Puerta del Mar, Cadiz, Spain